CLINICAL TRIAL: NCT04975555
Title: A Phase II Pilot Study to Evaluate the Role of Siltuximab in Treatment of Cytokine Release Syndrome (CRS) and Immune Effector Cell Associated Neurotoxicity (ICANS) Related to Chimeric Antigen Receptor T-Cell Therapy (CAR-T) in Hematological Malignancies
Brief Title: Study to Evaluate the Role of Siltuximab in Treatment of Cytokine Release Syndrome (CRS) and Immune Effector Cell Associated Neurotoxicity (ICANS) Related to CAR-T Cell Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Amitkumar Mehta, MD, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300007103
Record Dates: First submitted 2021-07-05; First posted 2021-07-23 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cytokine Release Syndrome; ICANS; Lymphoma, Non-Hodgkin; Multiple Myeloma; Acute Lymphoblastic Leukemia
Keywords: Siltuximab; Chimeric Antigen Receptor T-cell Therapy; Cytokine release syndrome; Immune effector Cell associated Neurotoxicity Syndrome; Lymphoma; Multiple Myeloma; Acute lymphoblastic Leukemia
MeSH Terms: conditions — Cytokine Release Syndrome; Lymphoma, Non-Hodgkin; Multiple Myeloma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma | interventions — siltuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Siltuximab (Experimental): Patients who experience CRS/ICANS will receive this treatment
  Interventions: Drug: Siltuximab

INTERVENTIONS:
Drug: Siltuximab — Siltuximab is administered at the dose of 11mg/kg via intravenous infusion over 1 hour. If no resolution of CRS is achieved then a repeat dose of siltuximab at the dose of 11mg/kg via intravenous infusion over 1 hour will be given.

SUMMARY:
This study will evaluate the use of siltuximab to decrease the severity of cytokine release syndrome (CRS) and immune effector cell-associated neurological syndrome (ICANS) in patients who will receive chimeric antigen receptor (CAR) T-cell therapy for the treatment of hematological malignancies.

DETAILED DESCRIPTION:
Patients eligible to receive CAR T-cell therapy for FDA-approved indications in hematological malignancies will be enrolled in this study on the day of CAR T-cell infusion. Patients will be followed until they develop grade 1 or higher CRS and/or ICANS. On developing these syndromes, siltuximab will be administered with close monitoring and follow-up for resolution of symptoms. If symptoms continue to worsen, then an additional dose of siltuximab will be given. If the symptoms leading to CRS do not resolve, then rescue tocilizumab will be administered. The study's primary endpoint is to assess the response rate of siltuximab in the resolution of CRS within 14 days. The study's secondary endpoint is to assess the response rate of siltuximab in the resolution of ICANS, the safety of siltuximab, and the overall response rate of CAR T-cell therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are planned to receive chimeric antigen receptor T-cell therapy as per the United States Food and Drug Agency (USFDA) approved indications for Diffuse large B-cell lymphoma (DLBCL), Mantle cell lymphoma (MCL), Follicular lymphoma (FL), Primary mediastinal large B-cell lymphoma (PMBCL), High grade B-cell lymphoma, DLBCL arising from follicular lymphoma, Multiple myeloma and B-cell precursor acute lymphoblastic leukemia
* Patients with hepatitis C virus (HCV) can be included if they have completed therapy for hepatitis C with undetectable HCV RNA viral load.
* Patients with Hepatitis B can be included if they are on suppressive therapy for hepatitis B infection and with no detectable viral load.
* Adequate organ function as defined below unless attributed to disease involvement.Acceptable window for assessing adequate organ function is 7 days to 30 days before planned CAR T-cell infusion with day 0 as the planned day of CAR T-cell infusion.Adequate liver function (bilirubin < 2mg/dL, aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) <3 x ULN), adequate kidney function (crcl > 30ml/min using Cockcroft-Gault, based on actual weight) and adequate hematological parameters (Absolute neutrophil count ≥ 1,000/µL, Hemoglobin > 8, Platelet Count ≥ 50,000/ µL)
* Patients able to tolerate washout periods for therapies prior to CAR T-cell infusion. Systemic therapy: Washout period is 2 weeks prior to CAR T-cell infusion. Radiation therapy: Washout period is 1 week prior to CAR T-cell infusion. Corticosteroids: The washout period is 5 days prior to CAR T-cell infusion.
* A negative urine pregnancy test is required within 1 week for all women of childbearing potential prior to enrolling on this trial.
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 4 months after infusion of siltuximab.
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner
* Willing and able to participate in all required evaluations and procedures in this study protocol including receiving intravenous administration of the investigational product and being admitted, when required, for at least 24 hours during investigational product administration.

Exclusion Criteria:

* Subjects requiring ongoing daily corticosteroid therapy at a dose of > 10 mg of prednisone per day (or equivalent). Pulsed corticosteroid use for disease control is acceptable.
* Active autoimmune disease requiring immunosuppressive therapy is excluded unless discussed with the principal investigator (PI)
* Pregnant women are excluded from this study.
* Evidence of ongoing systemic bacterial, or fungal or viral infection, except localized fungal infection of skin or nails.
* Patients with ongoing or past HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Participants with a complete response for cytokine release syndrome (CRS) | Baseline through 14 days
  Participants who achieve a resolution of CRS. Resolution of CRS is defined as absence of symptoms leading to diagnosis of CRS for 24 hours.

SECONDARY OUTCOMES:
Participants with a response for Immune effector Cell Associated Neurotoxicity Syndrome (ICANS) | Baseline through 28 days
  Participants who achieve a resolution or improvement in their ICANS. Complete response or partial response for ICANS is defined as either complete disappearance or decrease in the grade of severity as measured by ASTCT Consensus Grading for ICANS. The ASTCT grade is from 1 to 5 for ICANS with 1 being mild symptoms and 5 being severe symptoms.
Participants experiencing adverse events from Siltuximab | Baseline through 28 days
  All Adverse Events (AE's) will be reported and evaluated using National Cancer Institute's Common Terminology Criteria (CTCAE) v5.0.
Participants with response to CAR T-cell therapy | Baseline through day 90
  This will be measured by using specific criteria's for Lymphoma, Multiple Myeloma or Acute Lymphoblastic Leukemia (ALL) [Based on the patients diagnosis]

CONTACTS AND LOCATIONS:
Overall Officials: Amitkumar Mehta, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
To Be determined